CLINICAL TRIAL: NCT00917202
Title: Efficacy of Methylene Blue for Malaria Treatment in Adults of Burkina Faso: Proof of Principle Study in Semi-Immune Adults of Burkina Faso in the Frame of the A8
Brief Title: Efficacy of Methylene Blue for Malaria Treatment in Adults of Burkina Faso: Proof of Principle Study in Semi-Immune Adults of Burkina Faso in the Frame of the A8 Project of the SFB 544
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Other Study IDs: S-237/2007
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

ARMS (3):
- MB3 (Experimental): 3 days
  Interventions: Drug: Methylenblue
- MB5 (Experimental): 5 days
  Interventions: Drug: Methylenblue
- MB7 (Experimental)
  Interventions: Drug: Methylenblue

INTERVENTIONS:
Drug: Methylenblue

SUMMARY:
Design: Single-centre, controlled study in adults with uncomplicated falciparum malaria in the Nouna Health District, north-western Burkina Faso

Phase: Phase II

Objectives: The primary objective of this trial is to study the efficacy of different methylene blue regimens given to adults with uncomplicated falciparum malaria in an African area of high malaria transmission intensity.

Population: Male adults with uncomplicated malaria from Nouna town.

Sample size: N= 60 (n=20 for each group; three different dosing regimens of MB).

Treatment: The participants in the three different MB regimens will receive orally twice daily 390 mg MB (total daily dose 780mg) over 7,5 or 3 days respectively. Treatment with the five (three) day regimen will only start after all patients of the seven (five) days regimen have been followed up until day 3.

Endpoints: The primary endpoint is the adequate clinical and parasitological response (ACPR) rate on day 28. Secondary endpoints are the number of adverse events (AE) after drug intake until day 28, clinical and parasitological failure rates on day 14 and 28, changes in haemoglobin/haematocrit until day 28, and fever and parasite clearance time.

ELIGIBILITY:
Inclusion Criteria:

* Male adults (>17 years;<55 years)
* Uncomplicated malaria caused by P. falciparum
* Asexual parasites ≥ 1000/µl and ≤ 200 000/µl
* Axillary temperatures ≥ 37.5°C or history of fever during 48 hours
* Living in nouna Health District
* Informed consent

Exclusion Criteria:

* Complicated or severe malaria
* Any apparent significant disease
* Anaemia (haematocrit < 21%)
* Antimalarial treatment prior to inclusion (last three days)
* Increased creatinine blood levels

Ages: 17 Years to 55 Years | Sex: Male
Age Groups: Child, Adult

PRIMARY OUTCOMES:
Adequate clinical and parasitolgical response (ACPR) until D 28

SECONDARY OUTCOMES:
Early treatment failure (ETF) rate
Late clinical failure (LCF) rate at D14 and D28
Late parasitological failure (LPF) rate at D14 and D28
Fever clearance time
Parasite clearance time
Change in haematocrit after 2,3,7,14 and 28 days compared to baseline
Incidence of observed and self-reported non-serious adverse events over the 28 days observation period
Incidence of serious adverse events over the 28 days observation period
MB whole blood concentrations (trough concentrations) on day 3,5 or 7 compared to trough concentrations after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- Nouna Health District, Nouna, Burkina Faso